CLINICAL TRIAL: NCT01969747
Title: A 28-day Randomised, Placebo-controlled, Double-blind Parallel Group Phase IIa Trial to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Once Daily Oral Doses of 2.5 mg, 10 mg, and 25 mg Empagliflozin as Adjunctive to Insulin in Patients With Type 1 Diabetes Mellitus (EASE-2)
Brief Title: Empagliflozin add-on to Insulin in Type 1 Diabetes Mellitus Over 28 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.78; 2011-004354-25 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (4):
- Empagliflozin low (Experimental): Empagliflozin low once daily
  Interventions: Drug: Empagliflozin medium placebo; Drug: Empagliflozin high placebo; Drug: Empagliflozin low
- Empagliflozin medium (Experimental): Empagliflozin medium once daily
  Interventions: Drug: Empagliflozin low placebo; Drug: Empagliflozin high placebo; Drug: Empagliflozin medium
- Empagliflozin high (Experimental): Empagliflozin high once daily
  Interventions: Drug: Empagliflozin medium placebo; Drug: Empagliflozin low placebo; Drug: Empagliflozin high
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Empagliflozin low placebo; Drug: Empagliflozin high placebo; Drug: Empagliflozin medium placebo

INTERVENTIONS:
Drug: Empagliflozin medium placebo — Empagliflozin medium placebo
  Arms: Empagliflozin high
Drug: Empagliflozin low placebo — Empagliflozin low placebo
  Arms: Empagliflozin medium
Drug: Empagliflozin low placebo — Empagliflozin low placebo
  Arms: Placebo
Drug: Empagliflozin high placebo — Empagliflozin high placebo
  Arms: Empagliflozin medium
Drug: Empagliflozin medium — Empagliflozin medium
  Arms: Empagliflozin medium
Drug: Empagliflozin medium placebo — Empagliflozin medium placebo
  Arms: Empagliflozin low
Drug: Empagliflozin high placebo — Empagliflozin high placebo
  Arms: Empagliflozin low
Drug: Empagliflozin high placebo — Empagliflozin high placebo
  Arms: Placebo
Drug: Empagliflozin medium placebo — Empagliflozin medium placebo
  Arms: Placebo
Drug: Empagliflozin low placebo — Empagliflozin low placebo
  Arms: Empagliflozin high
Drug: Empagliflozin low — Empagliflozin low
  Arms: Empagliflozin low
Drug: Empagliflozin high — Empagliflozin high
  Arms: Empagliflozin high

SUMMARY:
Placebo-controlled, double blind (triple-dummy technique), randomised parallel design comparison of three oral doses (2.5 mg, 10 mg, and 25 mg) of empagliflozin in patients with T1DM as adjunctive therapy to insulin over 28 days. Patients will undergo a 14-day open-label placebo run-in period before randomisation. Background insulin therapy will be kept stable during the first 7 days of the treatment period and will be freely adjusted thereafter.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent
* Male or female patient receiving insulin for treatment of T1DM for at least 12 months
* C-peptide < 1.5 ng/mL
* Age 18 to 65 years
* HbA1c of 7.5% to 10.5%
* Multiple daily injections (MDI) of any type of insulin
* Willing to follow an established and individualized carbohydrate counting method and an insulin administration algorithm
* Body Mass Index of 18.5 to 35.0 kg/m2
* Estimated glomerular filtration rate 60 to 150 mL/min/1.73 m²
* Able and willing to perform study assessments according to investigator's judgement
* Compliance with trial drug administration 80% to 120% during run-in period
* Willing not to take any paracetamol containing drugs during the trial

Exclusion criteria:

* Acute symptomatic urinary tract infection or genital infection, chronic or recurrent cystitis
* History of type 2 diabetes mellitus, maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
* Pancreas, pancreatic islet cells or renal transplant recipient
* Type 1 diabetes mellitus treatment with any other antihyperglycaemic drug except insulin within last 3 months or history of clinically relevant hypersensitivity
* Occurrence of hypoglycaemia that required hospitalization or treatment by an emergency physician or paramedic within last 3 months
* Hypoglycaemia unawareness or frequent episodes of unexplained hypoglycaemia
* Occurrence of diabetic ketoacidosis that required hospitalization or treatment by an emergency physician or paramedic within last 12 months
* History of macrovascular disease including cardiovascular, cerebrovascular and peripheral artery disease
* Autonomic neuropathy with gastroparesis
* Brittle diabetes
* Liver disease
* Treatment with anti-obesity drugs, surgery or aggressive diet regimen leading to unstable body weight
* Treatment with systemic corticosteroids
* Change in dose of thyroid hormones within last 6 weeks or planned change or initiation of such a therapy
* Medical history of cancer or treatment for cancer in the last five years
* Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells
* Alcohol or drug abuse that would interfere with trial participation or any ongoing clinical condition that would jeopardize patient's or site personnel's safety or study compliance
* Intake of an investigational drug in another trial within last 30 days
* Not able to understand and comply with study requirements
* Pre-menopausal women who are nursing or pregnant or of child-bearing potential and are not practising an acceptable method of birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- 1245.78.43001 Boehringer Ingelheim Investigational Site, Graz, Austria
- 1245.78.49001 Boehringer Ingelheim Investigational Site, Neuss, Germany

REFERENCES:
- [Derived] Famulla S, Pieber TR, Eilbracht J, Neubacher D, Soleymanlou N, Woerle HJ, Broedl UC, Kaspers S. Glucose Exposure and Variability with Empagliflozin as Adjunct to Insulin in Patients with Type 1 Diabetes: Continuous Glucose Monitoring Data from a 4-Week, Randomized, Placebo-Controlled Trial (EASE-1). Diabetes Technol Ther. 2017 Jan;19(1):49-60. doi: 10.1089/dia.2016.0261. Epub 2016 Dec 8. PMID 27929674
- [Derived] Lamos EM, Younk LM, Davis SN. Empagliflozin, a sodium glucose co-transporter 2 inhibitor, in the treatment of type 1 diabetes. Expert Opin Investig Drugs. 2014 Jun;23(6):875-82. doi: 10.1517/13543784.2014.909407. Epub 2014 Apr 19. PMID 24746173

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet; oral administration once daily
- Empagliflozin 2.5 mg: Empagliflozin 2.5 mg tablet; oral administration once daily
- Empagliflozin 10 mg: Empagliflozin 10 mg tablet; oral administration once daily
- Empagliflozin 25 mg: Empagliflozin 25 mg tablet; oral administration once daily
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 19 | 19 | 19 | 18
Completed | 19 | 19 | 19 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all patients randomised, treated with at least one dose of study drug, had a baseline UGE (g/24 h) and a UGE (g/24 h) on Day 1 or Day 7.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 19 | 19 | 19 | 18 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (10.6) | 41.9 (12.4) | 39.6 (11.6) | 41.9 (9.7) | 41.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 8 | 22
  Male | 13 | 15 | 15 | 10 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24 h UGE (g/24 h) After Seven Days of Treatment With Empagliflozin 2.5 mg, 10 mg, or 25 mg, or Placebo
Description: Change of urinary glucose excretion (UGE) (g/24 h) from baseline (refers to the last measurement prior to the first intake of any randomised trial medication) after seven days of treatment with empagliflozin 2.5 mg, 10 mg, or 25 mg, or placebo.
  The treatment effect was estimated on the basis of the least square mean treatment difference at Day 7 extracted from the primary analysis model.
  The primary endpoint is exploratory.
Time Frame: baseline (Day -1) and 7 days after first drug administration (Day 7)
Population: Full analysis set (FAS): all patients randomised, treated with at least one dose of study drug, had a baseline UGE (g/24 h) and a UGE (g/24 h) on Day 1 or Day 7.
  The last observation carried forward (LOCF) approach was used as the primary method of imputation for missing data.
Measure: Mean (Standard Error); unit: g/24h
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 19 | 19 | 19 | 18
g/24h | -3.56 (4.27) | 72.45 (7.01) | 103.33 (6.68) | 101.79 (6.51)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 2.5 mg; Comparison of Empagliflozin 2.5 mg with Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean = 76.09, 95% CI 2-sided [58.60 to 93.59], Standard Error of Mean 8.77 — The model includes baseline UGE as linear covariate(s) and treatment as fixed effect(s)
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg; Comparison of Empagliflozin 10 mg with Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean = 106.39, 95% CI 2-sided [88.73 to 124.05], Standard Error of Mean 8.85 — The model includes baseline UGE as linear covariate(s) and treatment as fixed effect(s)
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg; Comparison of Empagliflozin 25 mg with Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean = 104.81, 95% CI 2-sided [86.88 to 122.74], Standard Error of Mean 8.99 — The model includes baseline UGE as linear covariate(s) and treatment as fixed effect(s)

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after last drug administration (Day 35)
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 17/19 | 17/19 | 15/19 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Empagliflozin 2.5 mg (N=19) | Empagliflozin 10 mg (N=19) | Empagliflozin 25 mg (N=18)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Empagliflozin 2.5 mg (N=19) | Empagliflozin 10 mg (N=19) | Empagliflozin 25 mg (N=18)
Nasopharyngitis (Infections and infestations) | 5 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 16 | 13 | 17
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 2 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.